CLINICAL TRIAL: NCT05433571
Title: Evaluation of Rotation With a Multifocal Toric Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6491
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-06

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (8):
- Myopes - Against the Rule Sequence 1 (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized to the Myope, against-the-rule-astigmatism, (LOW/HIGH DC) sequence and wear two different study lens designs one at a time bilaterally over 2 wear periods.
  Interventions: Device: Test Lens
- Myopes - Against the Rule Sequence 2 (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized to the Myope, against-the-rule-astigmatism, (HIGH/LOW DC) sequence and wear two different study lens designs one at a time bilaterally over 2 wear periods.
  Interventions: Device: Test Lens
- Myopes - With the Rule Sequence 1 (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized to the Myope, with-the-rule-astigmatism, (LOW/HIGH DC) sequence and wear two different study lens designs one at a time bilaterally over 2 wear periods.
  Interventions: Device: Test Lens
- Myopes - With the Rule Sequence 2 (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized to the Myope, with-the-rule-astigmatism, (HIGH/LOW DC) sequence and wear two different study lens designs one at a time bilaterally over 2 wear periods.
  Interventions: Device: Test Lens
- Hyperopes - Against the Rule Sequence 1 (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized to the Hyperope, against-the-rule-astigmatism, (LOW/HIGH DC) sequence and wear two different study lens designs one at a time bilaterally over 2 wear periods.
  Interventions: Device: Test Lens
- Hyperopes - Against the Rule Sequence 2 (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized to the Hyperope, against-the-rule-astigmatism, (HIGH/LOW DC) sequence and wear two different study lens designs one at time bilaterally over 2 wear periods.
  Interventions: Device: Test Lens
- Hyperope - With the Rule Sequence 1 (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized to the Hyperope, with-the-rule-astigmatism, (LOW/HIGH DC) sequence and wear two different study lens designs one at a time bilaterally over 2 wear periods.
  Interventions: Device: Test Lens
- Hyperope - With the Rule Sequence 2 (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized to the Hyperope, with-the-rule-astigmatism, (HIGH/LOW DC) sequence and wear two different study lens designs one at a time bilaterally over 2 wear periods.
  Interventions: Device: Test Lens

INTERVENTIONS:
Device: Test Lens — Multifocal Toric Contact Lenses manufactured in Senofilcon A (C3) material with UV/HEV filter

SUMMARY:
The study is a bilateral, single-masked, single-visit, non-dispensing 2x2 crossover study to confirm a finalized design of a prototype contact lens. There will be eight study lens types, however, each subject will only be randomized to receive two study lens types.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be at least 40 and not more than 70 years of age at the time of screening.
4. Own a wearable pair of spectacles with distance vision correction.
5. Be an adapted soft contact lens wearer in both eyes (i.e. has worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for the past four weeks).
6. Have distance spherical equivalent refraction in the range of either -1.00 D to -6.00 D or +1.00 to +6.00 D in each eye.
7. Have distance cylinder refraction in the range of -0.75 to - 2.50 D in each eye, with the axis being in the range of either 90 ± 30° or 180 ± 30°.
8. Have best corrected distance visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or lactating.
2. Have any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
3. Have any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens- Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
4. Use systemic medications that may interfere with contact lens wear or cause blurred vision. See section 9.1 for additional details regarding excluded systemic medications.
5. Currently use ocular medication with the exception of rewetting drops.
6. Have any known hypersensitivity or allergic reaction to single use preservative free rewetting drops, or sodium fluorescein.
7. Have had any previous ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
8. Have a history of amblyopia or strabismus.
9. Have a history of herpetic keratitis.
10. Have a history of irregular cornea.
11. Have a history of pathological dry eye.
12. Have participated in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
13. Be an employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
14. Have clinically significant (Grade 3 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
15. Have entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions.
16. Have any current ocular infection or inflammation.
17. Have any other ocular abnormality that may interfere with contact lens wear

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (5):
- United States (5):
  - Stam & Associates Eye Care, Jacksonville, Florida
  - Sabal Eye Care, Longwood, Florida
  - Maitland Vision Center - North Orlando Ave, Maitland, Florida
  - Center for Ophthalmic and Vision Research/Eye Associates of New York, Manhattan, New York
  - Tyler Eye Associates, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 102 subjects were enrolled in this study. Of those enrolled, all subjects were dispensed both lenses and completed the study. No subjects were discontinued.
Groups:
- Senofilcon A(C3) Toric Lens UV/HEV Filter(Low DC)/Senofilcon A(C3) Toric Lens UV/HEV Filter(High DC): Subjects randomized to this sequence received the Senofilcon A (C3) Multifocal Toric lens with UV/HEV filter (Low DC) during the first period and then received the Senofilcon A (C3) Multifocal Toric lens with UV/HEV filter (High DC) during the second period
- Senofilcon A(C3) Toric Lens UV/HEV Filter(High DC)/Senofilcon A(C3) Toric Lens UV/HEV Filter(Low DC): Senofilcon A (C3) Multifocal Toric lens with UV/HEV filter (High DC) during the first period and then received the Senofilcon A (C3) Multifocal Toric lens with UV/HEV filter (Low DC) during the second period
Period: Period 1
Arm/Group | Senofilcon A(C3) Toric Lens UV/HEV Filter(Low DC)/Senofilcon A(C3) Toric Lens UV/HEV Filter(High DC) | Senofilcon A(C3) Toric Lens UV/HEV Filter(High DC)/Senofilcon A(C3) Toric Lens UV/HEV Filter(Low DC)
Started | 53 | 49
Completed | 53 | 49
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Senofilcon A(C3) Toric Lens UV/HEV Filter(Low DC)/Senofilcon A(C3) Toric Lens UV/HEV Filter(High DC) | Senofilcon A(C3) Toric Lens UV/HEV Filter(High DC)/Senofilcon A(C3) Toric Lens UV/HEV Filter(Low DC)
Started | 53 | 49
Completed | 53 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed at least one study lens.
Groups:
- Total: Total Subjects
Arm/Group | Total
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black or African American | 6
  White | 93
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States: participants | 102

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes With Absolute Rotation ≤ 10 Degrees
Description: Absolute rotation was assessed for each subject eye using a slit lamp, at 1-, 3-, 7-, 15- and 25-minutes after lens insertion. However, absolute rotation at 15-minutes was the primary endpoint. Acceptable absolute rotation was dichotomized into a binary response where Y=1 if absolute rotation was less than or equal to 10 degrees and Y=0 otherwise (absolute rotation greater than 10 degrees). The proportion of eyes with absolute rotation less than or equal to 10 degrees was report for each lens.
Time Frame: 15-minutes post lens insertion
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion
Units Other Than Participants: Eyes
Groups:
- Senofilcon A (C3) Multifocal Toric Lens With UV/HEV Filter (Low DC): Subjects that wore the Test lens Senofilcon A (C3) Multifocal Toric lens with UV/HEV filter (Low DC) in either the first or second period of the study.
- Senofilcon A (C3) Multifocal Toric Lens With UV/HEV Filter (High DC): Subjects that wore the Senofilcon A (C3) Multifocal Toric lens with UV/HEV filter (High DC) in either the first or second period of the study.
Arm/Group | Senofilcon A (C3) Multifocal Toric Lens With UV/HEV Filter (Low DC) | Senofilcon A (C3) Multifocal Toric Lens With UV/HEV Filter (High DC)
Number analyzed (Participants) | 102 | 102
Number analyzed (Eyes) | 204 | 204
Proportion | 0.9167 | 0.8873
Statistical Analysis 1: Comparison: Senofilcon A (C3) Multifocal Toric Lens With UV/HEV Filter (Low DC); Test type: Superiority — Superiority was tested for Senofilcon A (C3) Multifocal Toric lens with UV/HEV filter (Low DC) and concluded if the lower limit of a 95% confidence interval was above 0.80; Bootstrapping Methods; bias adjusted confidence intervals; Mean Population Estimate = 0.917, 95% CI 2-sided [0.878 to 0.955], Standard Error of Mean 0.0194
Statistical Analysis 2: Comparison: Senofilcon A (C3) Multifocal Toric Lens With UV/HEV Filter (High DC); Test type: Superiority — Superiority was tested for Senofilcon A (C3) Multifocal Toric lens with UV/HEV filter (High DC) and concluded if the lower limit of a 95% confidence interval was above 0.80; Bootstrapping Methods; bias adjusted confidence intervals; Mean Population Estimate = 0.887, 95% CI 2-sided [0.845 to 0.930], Standard Error of Mean 0.0219

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 1-Day per Subject.
Description: All subjects dispensed at least 1 study lens.
Groups:
- Senofilcon A (C3) Multifocal Toric Lens With UV/HEV Filter (Low C): Subjects that wore the Test lens Senofilcon A (C3) Multifocal Toric lens with UV/HEV filter (Low DC) in either the first or second period of the study
Arm/Group | Senofilcon A (C3) Multifocal Toric Lens With UV/HEV Filter (Low C) | Senofilcon A (C3) Multifocal Toric Lens With UV/HEV Filter (High DC)
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/102
Other Adverse Events (participants affected / at risk) | 0/102 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT05433571/Prot_SAP_000.pdf